CLINICAL TRIAL: NCT01539408
Title: Sublingual Misoprostol Versus Standard Surgical Care for the Treatment of Incomplete Abortion
Brief Title: Sublingual Misoprostol Versus Standard Surgical Care for the Treatment of Incomplete Abortion in Nigeria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.2.3
Record Dates: First submitted 2012-02-16; First posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Incomplete Abortion
MeSH Terms: conditions — Abortion, Incomplete | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): 400 mcg of sublingual misoprostol in one dose
  Interventions: Drug: Misoprostol
- Manual vacuum aspiration (MVA) (Active Comparator): Standard surgical treatment (MVA)
  Interventions: Procedure: surgery Manual vacuum aspiration (MVA)

INTERVENTIONS:
Drug: Misoprostol — single dose of 400 mcg misoprostol administered sublingually
  Arms: Misoprostol
Procedure: surgery Manual vacuum aspiration (MVA) — standard surgical treatment
  Arms: Manual vacuum aspiration (MVA)

SUMMARY:
Women diagnosed with incomplete abortion in this health facility will be randomized to receive one of the following regimens: 400 mcg sublingual misoprostol in one dose or standard surgical treatment (MVA). The investigators hypothesize that treatment of incomplete abortion with misoprostol using 400 mcg administered sublingually will be as effective as surgical evacuation.

ELIGIBILITY:
Inclusion Criteria:

* no contraindications to misoprostol
* uterine size was not larger than 12 weeks
* there were no signs of severe infection
* haemodynamically stable
* in general good health
* willing to provide contact information

Exclusion Criteria:

* an IUD in place
* ectopic pregnancy
* aged below 18 years and had no accompanying adult to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Complete abortion without recourse to surgical intervention | follow up visit 7 days after initial treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Nigeria (2):
  - Adeoyo Maternity Hospital, Ibadan
  - University College Hospital, Ibadan, Ibadan

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352
- [Derived] Shochet T, Diop A, Gaye A, Nayama M, Sall AB, Bukola F, Blandine T, Abiola OM, Dao B, Olayinka O, Winikoff B. Sublingual misoprostol versus standard surgical care for treatment of incomplete abortion in five sub-Saharan African countries. BMC Pregnancy Childbirth. 2012 Nov 14;12:127. doi: 10.1186/1471-2393-12-127. PMID 23150927
- [Derived] Fawole AO, Diop A, Adeyanju AO, Aremu OT, Winikoff B. Misoprostol as first-line treatment for incomplete abortion at a secondary-level health facility in Nigeria. Int J Gynaecol Obstet. 2012 Nov;119(2):170-3. doi: 10.1016/j.ijgo.2012.06.012. Epub 2012 Aug 27. PMID 22935620